CLINICAL TRIAL: NCT01513148
Title: The Effect of Light Therapy on Superficial Radial Nerve Conduction Using a Clustered Array of Infrared Super Luminous and Red Light Emitting Diodes
Brief Title: Effects of Light Emitting Diode Irradiation on the Conduction Parameters of the Superficial Radial Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Todd Telemeco, Associate Professor, Shenandoah University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 06-750
Record Dates: First submitted 2012-01-09; First posted 2012-01-20 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Superluminous Light Diode Irradiation (Experimental): Application of super luminous diodes light irradiation over the superficial radial nerve
  Interventions: Device: Superluminous light diode
- Sham Superluminous Light Diode Irradiation (Placebo Comparator): Sham Superluminous Light Diode Irradiation over the Superficial Radial Nerve for the same time period as the intervention group
  Interventions: Device: Superluminous light diode

INTERVENTIONS:
Device: Superluminous light diode — 900W, 880nm, 1.6 J/cm2 for 30sec
  Other Names: Dynatronics Solaris Model 705

SUMMARY:
The introduction of light emitting diode (LED) devices as a novel treatment for pain relief in place of low-level laser warrants fundamental research on the effect of LED devices on one of the potential explanatory mechanisms: peripheral neurophysiology in vivo. A randomized controlled study will be conducted by measuring nerve conduction on the superficial radial nerve of healthy subjects (n=64). One baseline measurement and five post-irradiation recordings (2-min interval each) will be performed of the nerve conduction velocity (NCV) and peak latency (PL) and peak amplitude (PA). The experimental group (=32) will receive an irradiation of 2 J/cm2 with an infrared LED device (Dynatronics Solaris Model 705), while the placebo group will be treated by sham irradiation. The purpose of this study is to investigate the effects of LED light on the conduction velocity and amplitude of the superficial radial nerve.

ELIGIBILITY:
Inclusion Criteria:

* no history of neurological disease, polyneuropathy, peripheral neuropathy or cervical radiculopathy

Exclusion Criteria:

* positive findings during the clinical screening examination suggestive of an underlying neurological disease, polyneuropathy, peripheral neuropathy or cervical radiculopathy.
* a history of a neurological disease, polyneuropathy, peripheral neuropathy or cervical radiculopathy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Telemeco, PhD, Principal Investigator — Shenandoah University
Locations (1):
- Shenandoah University Divsion of Physical Therapy, Winchester, Virginia, United States

REFERENCES:
- [Background] Greathouse DG, Currier DP, Gilmore RL. Effects of clinical infrared laser on superficial radial nerve conduction. Phys Ther. 1985 Aug;65(8):1184-7. doi: 10.1093/ptj/65.8.1184. PMID 4023064
- [Background] Downie AW, Scott TR. An improved technique for radial nerve conduction studies. J Neurol Neurosurg Psychiatry. 1967 Aug;30(4):332-6. doi: 10.1136/jnnp.30.4.332. No abstract available. PMID 4293407
- [Background] Snyder-Mackler L, Bork CE. Effect of helium-neon laser irradiation on peripheral sensory nerve latency. Phys Ther. 1988 Feb;68(2):223-5. doi: 10.1093/ptj/68.2.223. PMID 3340661

RESULTS

PARTICIPANT FLOW:
Groups:
- Light Therapy: Application of super luminous diodes light irradiation over the superficial radial nerve
- Sham Irradiation: Sham Irradiation over the Superficial Radial Nerve for the same time period as the intervention group
Period: Overall Study
Arm/Group | Light Therapy | Sham Irradiation
Started | 16 | 16
Completed | 14 | 14
Not Completed | 2 | 2
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Light Therapy | Sham Irradiation | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.5 (2.1) | 25.5 (3.9) | 24.7 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Nerve Conduction Velocity (Meters Per Second)
Description: Change in nerve conduction velocity (m/s) from pre-treatment to 0 minute (immediately after treatment), and at 2 min intervals after treatment until 10 minutes post treatment occurs. Calculated difference scores at each time point = nerve conduction velocity (NCV) - baseline NCV. A positive variance represented an increase from baseline and is interpreted as being an increase or faster velocity.
Time Frame: pre-treatment, 0 min, 2 min, 4 min, 6 min, 8 min and 10 min after treatment
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Light NCV Pretreatment: NCV at baseline, before the application of super luminous diodes light irradiation over the superficial radial nerve
- Light NCV Time 0: NCV at time 0, immediately following the application of super luminous diodes light irradiation over the superficial radial nerve
- Light NCV Time 2: NCV 2 minutes following the application of super luminous diodes light irradiation over the superficial radial nerve
- Light NCV Time 4: NCV 4 minutes following the application of super luminous diodes light irradiation over the superficial radial nerve
- Light NCV Time 6: NCV 6 minutes following the application of super luminous diodes light irradiation over the superficial radial nerve
- Light NCV Time 8: NCV 8 minutes following the application of super luminous diodes light irradiation over the superficial radial nerve
- Light NCV Time 10: NCV 10 minutes following the application of super luminous diodes light irradiation over the superficial radial nerve
- Sham NCV Pretreatment: NCV at baseline, before the application of sham superluminous diodes light irradiation over the superficial radial nerve
- Sham NCV Time 0: NCV immediately (Time 0) following the application of superluminous diodes light irradiation over the superficial radial nerve
- Sham NCV Time 2: NCV 2 minutes following the application of sham superluminous diodes light irradiation over the superficial radial nerve
- Sham NCV Time 4: NCV 4 minutes following the application of sham superluminous diodes light irradiation over the superficial radial nerve
- Sham NCV Time 6: NCV 6 minutes following the application of sham superluminous diodes light irradiation over the superficial radial nerve
- Sham NCV Time 8: NCV 8 minutes following the application of sham superluminous diodes light irradiation over the superficial radial nerve
- Sham NCV Time 10: NCV 10 minutes following the application of sham superluminous diodes light irradiation over the superficial radial nerve
Arm/Group | Light NCV Pretreatment | Light NCV Time 0 | Light NCV Time 2 | Light NCV Time 4 | Light NCV Time 6 | Light NCV Time 8 | Light NCV Time 10 | Sham NCV Pretreatment | Sham NCV Time 0 | Sham NCV Time 2 | Sham NCV Time 4 | Sham NCV Time 6 | Sham NCV Time 8 | Sham NCV Time 10
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14
m/s | 0.000 (0.000) | -0.358 (1.200) | 0.447 (1.616) | 0.147 (1.785) | -0.041 (1.741) | 0.280 (1.801) | 0.100 (2.117) | 0.000 (0.000) | 0.151 (1.251) | -0.004 (1.386) | 0.447 (1.616) | 1.116 (1.530) | 0.521 (1.652) | 0.675 (2.012)

2. Secondary Outcome: Negative Peak Latency (Milliseconds)
Description: Change in negative peak latency (ms) from pre-treatment to 0 minute (immediately after treatment), and at 2 min intervals after treatment until 10 minutes post treatment occurs. Calculated difference scores at each time period = negative peak latency NPL - baseline NPL. A positive variance can be interpreted as being increase from baseline or a prolonged or slowed NPL.
Time Frame: pre-treatment, 0 min, 2 min, 4 min, 6 min, 8 min and 10 min after treatment
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Light NPL Pre-treatment: NPL for treatment group (Superluminous diode light therapy) at baseline (pre-treatment)
- Light NPL Time 0: NPL for treatment group (Superluminous diode light therapy) at time 0 minutes
- Light NPL Time 2: NPL for treatment group (Superluminous diode light therapy) at time 2 minutes
- Light NPL Time 4: NPL for treatment group (Superluminous diode light therapy) at time 4 minutes
- Light NPL Time 6: NPL for treatment group (Superluminous diode light therapy) at time 6 minutes
- Light NPL Time 8: NPL for treatment group (Superluminous diode light therapy) at time 8 minutes
- Light NPL Time 10: NPL for treatment group (Superluminous diode light therapy) at time 10 minutes
- Sham NPL Time 0: NPL for Sham treatment group (Sham Superluminous diode light therapy) at time 0 minutes
- Sham NPL Time 2: NPL for Sham treatment group (Sham Superluminous diode light therapy) at time 2 minutes
- Sham NPL Time 4: NPL for Sham treatment group (Sham Superluminous diode light therapy) at time 4 minutes
- Sham NPL Time 6: NPL for Sham treatment group (Sham Superluminous diode light therapy) at time 6 minutes
- Sham NPL Time 8: NPL for Sham treatment group (Sham Superluminous diode light therapy) at time 8 minutes
- Sham NPL Time 10: NPL for Sham treatment group (Sham Superluminous diode light therapy) at time 10 minutes
- Sham NPL Pretreatment: NPL for Sham treatment group (Sham Superluminous diode light therapy) at baseline (pretreatment)
Arm/Group | Light NPL Pre-treatment | Light NPL Time 0 | Light NPL Time 2 | Light NPL Time 4 | Light NPL Time 6 | Light NPL Time 8 | Light NPL Time 10 | Sham NPL Time 0 | Sham NPL Time 2 | Sham NPL Time 4 | Sham NPL Time 6 | Sham NPL Time 8 | Sham NPL Time 10 | Sham NPL Pretreatment
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14
ms | 0.000 (0.000) | 0.414 (0.429) | 0.007 (0.070) | -0.007 (0.080) | 0 (0.755) | -0.014 (0.083) | -0.007 (0.096) | -0.007 (0.059) | 0.000 (0.065) | -0.021 (0.077) | -0.050 (0.073) | -0.021 (0.077) | -0.028 (0.096) | 0 (0)

3. Secondary Outcome: Temperature (Degrees C)
Description: Change in superficial skin temperature (degrees C) from pre-treatment to 0 minute (immediately after treatment), and at 2 min intervals after treatment until 10 minutes post treatment occurs. Calculated difference scores at each time point = Temperature - Temperature at baseline. A positive variance int his calculation can be interpreted as being an increase from baseline or an increase in skin temperature
Time Frame: pre-treatment, 0 min, 2 min, 4 min, 6 min, 8 min and 10 min after treatment
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Groups:
- Light Temp Pretreatment: Temperature prior to the application of super luminous diodes light irradiation over the superficial radial nerve
- Light Temp Time 0: Temperature immediately following the application of superluminous diodes light irradiation over the superficial radial nerve
- Light Temp Time 2; Sham Temp Time 2: Temperature 2 minutes following the application of superluminous diodes light irradiation over the superficial radial nerve
- Light Temp Time 4; Sham Temp Time 4: Temperature 4 minutes following the application of superluminous diodes light irradiation over the superficial radial nerve
- Light Temp Time 6; Sham Temp Time 6: Temperature 6 minutes following the application of superluminous diodes light irradiation over the superficial radial nerve
- Light Temp Time 8; Sham Temp Time 8: Temperature 8 minutes following the application of superluminous diodes light irradiation over the superficial radial nerve
- Light Temp Time 10; Sham Temp Time 10: Temperature 10 minutes following the application of superluminous diodes light irradiation over the superficial radial nerve
- Sham Temp Pretreatment: Temperature prior to the application of sham super luminous diodes light irradiation over the superficial radial nerve
- Sham Temp Time 0: Temperature immediately following the application of sham superluminous diodes light irradiation over the superficial radial nerve
Arm/Group | Light Temp Pretreatment | Light Temp Time 0 | Light Temp Time 2 | Light Temp Time 4 | Light Temp Time 6 | Light Temp Time 8 | Light Temp Time 10 | Sham Temp Pretreatment | Sham Temp Time 0 | Sham Temp Time 2 | Sham Temp Time 4 | Sham Temp Time 6 | Sham Temp Time 8 | Sham Temp Time 10
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14
Degrees Celsius | 0.000 (0.000) | 0.414 (0.429) | 0.993 (0.626) | 0.686 (1.210) | 0.757 (1.336) | 0.786 (1.341) | 0.778 (1.432) | 0.000 (0.000) | 0.814 (0.662) | 1.021 (0.591) | 0.993 (0.626) | 1.007 (0.796) | 0.928 (0.820) | 0.878 (0.847)

ADVERSE EVENTS:
Arm/Group | Light Therapy | Sham Irradiation
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
4 subjects were terminated early in the project, two from the light therapy group and two from the sham therapy group. All cases, we were unable to achieve an appropriate baseline temperature of 30 degrees celsius to allow continued participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes